CLINICAL TRIAL: NCT03034057
Title: PHASE IV OPEN LABEL SINGLE GROUP ONE YEAR STUDY OF HOME SELF-INJECTION WITH SAYANA (REGISTERED) PRESS IN ADULT WOMEN OF REPRODUCTIVE AGE - A PRAGMATIC CLINICAL TRIAL
Brief Title: Sayana Press UK Self-Injection Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A6791040; 2017-000051-13 (EudraCT Number)
Record Dates: First submitted 2017-01-24; First posted 2017-01-27 (Estimated); Results first posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-09

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sayana press (Other): single arm
  Interventions: Drug: Sayana Press

INTERVENTIONS:
Drug: Sayana Press — Sayana Press in the Uniject injection system

SUMMARY:
A one-year evaluation of Sayana Press self injection in women of reproductive age in the United Kingdom (UK).

ELIGIBILITY:
Inclusion Criteria:

* women aged 18 to 45 years of age who are willing to attempt Sayana Press self-injection at home;
* women who are likely to be successful on a DMPA self-injection program, based on the opinion of the investigator;
* not planning to move out of the area for at least 12 months;
* willing to be contacted by the clinical staff at work or at home;
* evidence of a personally signed and dated Informed Consent Document (ICD) indicating that the subject has been informed of all pertinent aspects of the study;
* subjects who are willing and able to comply with scheduled visits, treatment plan and other study procedures

Exclusion Criteria:

* a pre-existing medical condition that would interfere with participation in the study or pose a risk to the subject, including hypersensitivity to MPA or any constituents of Sayana Press;
* known or suspected malignancy of genital organs;
* known or suspected malignancy of the breast;
* history of cerebrovascular disease
* metabolic bone disease
* a contraindication to DMPA (UK Medical Eligibility Criteria Category 3 or 4) such as:
* Multiple risk factors for cardiovascular disease (e.g. older age, smoking, diabetes, obesity, hypertension)
* current and history of ischaemic heart disease;
* stroke (history of cerebrovascular accident, including transient ischaemic attack);
* unexplained vaginal bleeding;
* current or history of breast cancer;
* diabetic nephropathy, neuropathy, retinopathy or other diabetic vascular disease;
* severe (decompensated) liver cirrhosis;
* hepatocellular adenoma;
* hepatoma;
* Systemic Lupus Erythematosus (positive or unknown antiphospholipid antibodies; severe thrombocytopenia;
* subjects who are investigational centre staff members directly involved in the conduct of the study and their family members, centre staff members otherwise supervised by the investigator, or subjects who are Pfizer employees involved in the conduct of the study;
* participation in other studies involving investigational drug(s) within 30 days prior to study entry and/or during study participation;
* patients who plan to get pregnant within two years of study;
* breastfeeding and pregnant subjects;
* other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgement of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 169 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (26):
- United Kingdom (26):
  - Fowey Clinical Research Office, Fowey, Cornwall
  - Fowey River Practice, Fowey, Cornwall
  - Brannel Surgery, St Austell, Cornwall
  - Rame Medical Ltd, Penntorr Health, Torpoint, Cornwall
  - Rame Medical Ltd, Torpoint, Cornwall
  - Knowle House Surgery, Plymouth, Devon
  - NHS Ayrshire & Arran, University Hospital Crosshouse, Kilmarnock, EAST Ayrshire
  - Trafalgar Medical Group Practice, Southsea, Hampshire
  - NHS Highland Clinical Research Facility, Inverness, Highland
  - Kent Community Health NHS Foundation Trust, Canterbury, KENT
  - Kent Community Health NHS Foundation Trust, Chatham, KENT
  - Southport & Ormskirk Hospital NHS Trust, The May Logan Healthy Living Centre, Liverpool, Merseyside
  - Southport & Ormskirk Hospital NHS Trust, Liverpool, Merseyside
  - NHS Lothian, Chalmers Sexual Health Centre, Edinburgh, Midlothian
  - NHS Ayrshire & Arran, Ayrshire Central Hospital, Irvine, North Ayrshire
  - Pickering Medical Practice, Pickering, North Yorkshire
  - St Chad's Surgery, Radstock, Somerset
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, TYNE and WEAR
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, WEST Midlands
  - Eve Hill Medical Practice, Dudley, WEST Midlands
  - Bradford on Avon Health Centre, Bradford-on-Avon, Wiltshire
  - Hathaway Medical Centre, Chippenham, Wiltshire
  - Trowbridge Health Centre, Trowbridge, Wiltshire
  - Westbury Group Practice, Westbury, Wiltshire
  - CPS Research, Glasgow
  - Homerton University Hospital NHS Foundation Trust, Homerton, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A6791040

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 169 adult women participants of reproductive age (18 to 45 years) were enrolled in the study.
Groups:
- Sayana Press: Following product use education and a supervised initial self-injection at the baseline visit, participants self-injected Sayana Press in the home setting every 3 months (at Month 3, Month 6 and Month 9) and returned for a final study visit at Month 12.
Period: Overall Study
Arm/Group | Sayana Press
Started | 169
Completed | 114
Not Completed | 55
Not completed — Withdrawal by Subject | 10
Not completed — Protocol Violation | 1
Not completed — Not defined | 2
Not completed — Lost to Follow-up | 19
Not completed — Adverse Event | 22
Not completed — Medication error without associated AE | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who enrolled into the study.
Arm/Group | Sayana Press
Number analyzed (Participants) | 169
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.1 (7.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 154
  Unknown or Not Reported | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 163
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Successful Self-Injections Performed of All Attempts at Home on Schedule (Full Analysis Set)
Description: Each participant had a maximum of 3 home self-injections, each of which was defined as a success or failure. A success was defined as a home self-injection that was successfully performed by the participant at home and on schedule (13 week interval +/- 1 week) where all attempts were included in the denominator. If the participant attempted but was unable to administer the self-injection at home and had it performed instead at the clinic, then these were classed as failures. This outcome measure was analyzed by generalized estimating equation (GEE) model using participant as the clustering variable. The GEE model used the logit link and contained an intercept term. The 95% confidence interval (CI) for the intercept was transformed to a 95% CI for the self-injection success rate.
Time Frame: Up to 1 year
Population: The analysis population included participants who enrolled into the study.
Measure: Number (95% Confidence Interval); unit: Percentage of all attempts at home
Arm/Group | Sayana Press
Number analyzed (Participants) | 169
Percentage of all attempts at home | 88.8 [85.1 to 91.6]

2. Primary Outcome: Percentage of Successful Self-Injections Performed of All Attempts at Home on Schedule (Sensitivity Analysis)
Description: Each participant had a maximum of 3 home self-injections, each of which was defined as a success or failure. A success was defined as a home self-injection that was successfully performed by the participant at home and on schedule (13 week interval +/- 1 week) where all attempts were included in the denominator. If the participant attempted but was unable to administer the self-injection at home and had it performed instead at the clinic, then these were classed as failures. This outcome measure was analyzed by GEE model using participant as the clustering variable. The GEE model used the logit link and contained an intercept term. The 95% CI for the intercept was transformed to a 95% CI for the self-injection success rate. The sensitivity analysis was conducted to eliminate the data from the discontinued site due to ongoing Good Clinical Practice (GCP) violations.
Time Frame: Up to 1 year
Population: The analysis population included participants who enrolled into the study. Participants at sites which required closure during study due to GCP violations were excluded from the analysis population.
Measure: Number (95% Confidence Interval); unit: Percentage of all attempts at home
Arm/Group | Sayana Press
Number analyzed (Participants) | 164
Percentage of all attempts at home | 89.3 [85.6 to 92.1]

3. Secondary Outcome: Continuation Rate for the Method (Self-injection With Sayana Press) at 1 Year
Description: Continuation rate for the method at 1 year equals: ([the number of participants who received all 4 injections and had not discontinued by 12 months] / [total number of participants in the study]) *100%. A 95% CI was calculated along with the continuation rate using normal approximation to the binominal.
Time Frame: 1 year
Population: The analysis population included participants who enrolled into the study.
Measure: Number (95% Confidence Interval); unit: Percentage of total participants
Arm/Group | Sayana Press
Number analyzed (Participants) | 169
Percentage of total participants | 67.5 [59.8 to 74.5]

ADVERSE EVENTS:
Time Frame: Up to 1 year
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Sayana Press
All-Cause Mortality (participants affected / at risk) | 0/169
Serious Adverse Events (participants affected / at risk) | 5/169
Other Adverse Events (participants affected / at risk) | 60/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sayana Press (N=169)
Food poisoning (Gastrointestinal disorders) | 1 (1)
Mastitis (Infections and infestations) | 1 (1)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sayana Press (N=169)
Injection site bruising (General disorders) | 22 (25)
Injection site mass (General disorders) | 9 (9)
Injection site pain (General disorders) | 11 (12)
Depression (Psychiatric disorders) | 13 (13)
Vaginal haemorrhage (Reproductive system and breast disorders) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/57/NCT03034057/SAP_000.pdf
  • Study Protocol (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/57/NCT03034057/Prot_001.pdf